CLINICAL TRIAL: NCT03341858
Title: STRONG Kids 2: A Cells-to-Society Approach to Nutrition in Early Childhood
Acronym: SK2
Status: Active, not recruiting | Type: Observational
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: National Dairy Council (Other); The Gerber Foundation (Other); National Institutes of Health (NIH) (NIH); United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 13448
Record Dates: First submitted 2017-10-12; First posted 2017-11-14 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Child Obesity; Child, Only
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological and genetic sampling: Stool samples from infant and A stool sample from the mother will also be provided at the 6week home visit. A saliva sample will be collected at the 6 week home visit from both the mother and infant and again from the child at 4 years of age. A trained researcher will swab each participant's mouth and collect a small sample using a non-invasive technique. In order to more accurately assess the dietary intake of breast-fed and formula-fed infants we will be requesting a sample of the mother's breastmilk or the formula that she is feeding her infant at 6 weeks of age. The concentrations of nutrient and bioactive components in the breastmilk or formula will be analyzed. BREASTMILK SAMPLE: Breastfeeding mothers will be asked to provide a breast milk sample representative of the milk provided in the 24 hours prior to the fecal sample collection at 6 weeks postpartum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention-strictly observational

SUMMARY:
STRONG Kids 2: A Cells to Society Approach to Nutrition

Overview Using a cells-to-society approach to nutrition, this transdisciplinary project will provide unique insights into how individual biology interacts with the family environment to promote healthy eating habits in young children. It is one of the first studies to take a longitudinal look at the habits, including milk and dairy consumption, from birth. STRONG Kids 2 is built upon previous research from STRONG Kids 1 with preschool-aged children, documenting the relationship among genetic, child, and family factors in predicting BMI and dietary habits. The study sample includes 450 infants and their families located in small urban communities in central Illinois. Biological samples and height and weight measurements from infants and toddlers are collected at 6 weeks, 3, 12, 18 months and 2, 3, 4, 5, 6, 7 and 8 years. Mothers are surveyed about weaning, dietary habits, household routines, children's emotions, feeding styles, and milk and dairy consumption. Additional measures such as maternal height and weight are also being collected.

DETAILED DESCRIPTION:
Despite increased public awareness, there has been little progress over the past 2 decades in stemming the tide of childhood obesity in the U.S. Recent projections indicate that by 2030, at least 42% of American adults will be obese and 11% will be categorized as severely obese.Unfortunately, high rates of obesity begin in early childhood. According to the most recent estimates of obesity prevalence in U.S. children, 26.7% of 2-5 year-olds were overweight (>85th BMI percentile) and 12.1% were considered obese (>95th BMI percentile). Epidemiological data show that overweight and obesity during early childhood tracks into later childhood, adolescence, and adulthood.The persistence of unhealthy weight from early childhood into later years is multi factorial involving biological and behavioral facets, which may explain, in part, the relatively poor success of weight loss programs for children and adolescents.

The Synergistic Theory and Research on Obesity and Nutrition Group (STRONG) Kids Program (SKP) at the University of Illinois Urbana-Champaign is a well-established interdisciplinary research and education program aimed at identifying the multiple factors that contribute to unhealthy weight gain in preschool age (2-5 year-old) children. The team incorporates a "cells-to-society" approach, recognizing that biological and socio-environmental factors interact to affect eating and physical activity behaviors. The purpose of this project is to expand the STRONG Kids Program and launch a birth cohort study to examine the impact of food, milk, and dairy product consumption on weight trajectory from birth to five years of age. Due to the multidisciplinary expertise of our research team we will also examine the contributions of biological and environmental factors to the development of dietary habits, diet quality and the child's growth trajectory. The research team capitalize on emerging scientific findings that demonstrate that variability in individual biology(genetics), child self-regulation (e.g., inhibitory control), and family household characteristics (e.g., routines) make significant contributions to the development of satiety and food preferences during early childhood. This innovative longitudinal study will be the first of its kind to evaluate the composition of the gut microbiota over time and its potential impact on the self-regulatory personality characteristics in young children known to affect food preferences. Further, the research team will use well-established protocols to assess maternal and household characteristics known to promote healthy eating patterns to determine the intersection of child biological functioning and the introduction of solid foods, including milk and dairy foods, during the weaning period and their effects on weight trajectory up to three years of age.

The STRONG Kids Program 2 (SKP2), will recruit a cohort sample of 400 infants and their families into a comprehensive five-year longitudinal study that will be unique by its theory-driven integration of genetics, nutrition, child development and family science. This comprehensive approach will allow for a greater understanding of how dietary habits are established during the first five years of life and contribute to healthy weight. The team will collect biological samples (saliva and stool specimens) and height,weight from infants and toddlers at 1 and 6 weeks and 3 months, after the introduction of solid foods, 12, 18 months and 2, 3 , 4, 5, 6, 7 and 8 years postpartum.

Concordantly we will survey mothers about weaning, dietary habits, household routines, child self-regulation, feeding practices and styles, and maternal height and weight. This comprehensive approach is based on our first phase of STRONG Kids research (SKP1) with preschool age children, which has documented the relationship among child and family factors in predicting BMI and dietary habits. To date, there is scant evidence-based information on how parents make decisions to introduce new foods during the weaning period and the effects of different food types on child weight from birth to the early years. Specifically, there is a glaring absence of scientific information on the contribution that individual biology plays in positively interacting with milk and cultured dairy products(e.g, cheese, yogurt) as initial foods introduced during the weaning period and their contribution to sustaining healthy weight during the preschool years. This is likely to be a complex interaction among the child's biological make-up, temperament and response to satiety, the parent's feeding practices and styles, availability of food resources, and the feeding policies in place once the child is enrolled in child care. The STRONG Kids team has the expertise to address these multiple influences and can provide a fresh comprehensive approach to the study of food consumption and weight gain during the early years.

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

* preterm delivery
* non-singleton birth
* Down Syndrome
* Cleft palate
* Cystic Fibrosis
* Phenylketonuria [PKU]or other inborn errors of metabolism,
* a congenital heart condition that affects feeding,
* gene defects or hormone deficiencies that would affect growth.
* If an infant is born with any other rare defect not listed there, they will also be excluded from participation.

Ages: 0 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We will use enrollment of pregnant women recruited through three area hospitals and two clinics in the Champaign County region.Participants will be recruited in their last trimester of pregnancy in cooperation with OB/GYN and Family Practice Physicians at at Francis Nelson and Carle Foundation Hospital (Champaign), Christie Clinic (Champaign), Decatur Memorial Hospital (Decatur, IL), Provena United Samaritans Medical Center and Danville Polyclinic(Danville, IL). These recruitment sites will provide an adequate sample base to recruit 440 families.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2013-05-10 (Actual); Primary Completion 2027-08-20 (Estimated); Study Completion 2027-08-20 (Estimated)

PRIMARY OUTCOMES:
SK2 recruitment | Years 1-3
  Recruit 440 families (increased by 10% to retain cohort of 400 over time should budget permit)
Identify relationship between gut microbiota, weaning practices, and early milk consumption patterns | Years 1-12
  Identify relationship between gut microbiota, weaning practices, and early milk consumption patterns
Identify relationship between individual biology, family factors, and toddler food and dairy consumption | Years 1-12
  Identify relationship between individual biology, family factors, and toddler food and dairy consumption

CONTACTS AND LOCATIONS:
Overall Officials: Sharon M Donovan, PhD, Principal Investigator — University of Illinois Urbana Champaign; Barbara H Fiese, PhD, Principal Investigator — University of Illinois Urbana Champaign

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McMath AL, Iwinski S, Shen S, Bost KF, Donovan SM, Khan NA. Adherence to Screen Time and Physical Activity Guidelines is Associated with Executive Function in US Toddlers Participating in the STRONG Kids 2 Birth Cohort Study. J Pediatr. 2023 Jan;252:22-30.e6. doi: 10.1016/j.jpeds.2022.08.026. Epub 2022 Aug 24. PMID 36027980
- [Derived] Fiese BH, Musaad S, Bost KK, McBride BA, Lee SY, Teran-Garcia M, Donovan SM. The STRONG Kids 2 Birth Cohort Study: A Cell-to-Society Approach to Dietary Habits and Weight Trajectories across the First 5 Years of Life. Curr Dev Nutr. 2019 Jan 18;3(3):nzz007. doi: 10.1093/cdn/nzz007. eCollection 2019 Mar. PMID 30882062